CLINICAL TRIAL: NCT06146036
Title: A Comparison of the Acute Effects of Two ''Exercise Snacking'' Modalities on Glycemic Control in Overweight Patients With Type 2 Diabetes
Brief Title: Effects of Different ''Exercise Snacking'' Modalities on Glycemic Control in Patients With Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nis (Other)
Responsible Party: Principal Investigator, Anja Lazić, Junior Researcher, University of Nis
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: To snack or not to snack
Record Dates: First submitted 2023-11-13; First posted 2023-11-24 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Diabetes Mellitus, Type 2; Overweight or Obesity
Keywords: exercise, high intensity, diabetes melitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight; Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HIIT snacks (Experimental): 3 x 6×1 minute cycling intervals at 90% at HRmax
  Interventions: Behavioral: HIIT snacks
- Sprint snaks (Experimental): 3×20-second 'all-out' cycling with 1-4 hours recovery between sprints
  Interventions: Behavioral: Sprint snacks
- Control (Experimental): No exercise. Rest.
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: HIIT snacks — Cycling Exercise. 3 times per day 6 x 1 min at approximately 85-95% of HRmax
  Arms: HIIT snacks
Behavioral: Sprint snacks — Cycling Exercise. 3 times per day one ''all out'' sprint
  Arms: Sprint snaks
Other: Control — No exercise, sedentary.
  Arms: Control

SUMMARY:
Patients with type 2 diabetes (T2DM) face an increased risk of obesity, hypertension, and hyperglycemia, attributed to impaired cardiorespiratory fitness, elevated Hb1AC levels, and impaired lipid status. Therefore, effective prevention of complications and T2DM-related diseases is crucial for increasing the life expectancy of T2DM patients. Regular exercise plays a crucial role in the prevention and management of diabetes and its associated complications. However, most T2DM patients are not engaged in exercise. The most common causes are a lack of time, monotonous training patterns, and the severe exhaustion patients experience after recently developed and effective HIIT and SIT programs. Therefore, recent studies have explored the concept of "exercise snacking" (brief isolated bouts (< 1 min) of intense exercise spread throughout the day

) as a promising strategy to improve glycemic control, functional capacity, and cardiometabolic health among clinical and healthy populations. However, the type, intensity, and volume of exercise bouts that result in the best improvement are unknown. Therefore, we hypothesize that these exercise modalities may also acutely improve glycaemic control in sedentary overweight patients with T2DM.

1. This study will examine the acute impact of two modalities of ''Exercise Snacking'', compared with a no-exercise control (CON), on glycemic control and blood pressure
2. Compare the acute effects of two ''Exercise Snacking'' modalities
3. Collect data on individuals' perceptions of each workout mode using measures of Rate of Perceived Exertion (RPE), enjoyment, affect, and adverse events

DETAILED DESCRIPTION:
A randomized crossover design will be used for the acute effects study.

Prior to the experimental protocols, participants will be asked to come to the lab on four separate days, which will be scheduled to meet individual schedules.

Day one An electrocardiography stress test (ECG) test will be performed to assess if participants could enroll in the study. The test will be conducted, monitored, and reviewed by a Cardiologist and written approval will be necessary for further inclusion in the study. Moreover, during the first visit a continuous glucose monitoring (iCGM) device - will be inserted on the participant's non-dominant upper arm according to the manual guidelines. The accuracy of the iCGM devices will be validated using capillary vs interstitial iCGM measurements.

Day two The participants will be tested for anthropometric characteristics (height), and body composition. This procedure is necessary to determine the BMI most validly. All tests will be conducted in the laboratory of the Faculty of Sports and Physical Education.

Day three The maximal incremental test on the cycle ergometer will be used to determine the cardiorespiratory fitness level (VO2max, VO2peak) as well as the resting heart rate (HRrest), maximum HR (HRmax), and HR recovery (HRRTEST). These parameters, primarily HRmax will be crucial when implementing the intensity of the session which will not be done in an ''all effort'' manner. Participants will be familiarized with wearing the heart rate monitors and using the rating of perceived exertion scale (RPE) too. Briefly, after a 5-minute warm-up at 50 W, the intensity will be increased by 15 W/min until the tempo can no longer be maintained at 50 rpm. Cardiorespiratory fitness will be measured using an online gas analysis system (Cosmed Quark; CPET, Rome, Italy), VO2peak will be determined as the highest ten-breath rolling average and accepted if two or more of the following criteria were met: (1) voluntary exhaustion, (2) a plateau in VO2 despite increasing intensity; (3) maximal heart rate within 10 beats of the age-predicted maximum. This protocol already has been used in patients with T2DM.

Day four On the fourth day, the familiarization process will be conducted. Briefly, participants will be given the opportunity to try on the exercise sessions that we will use in the main protocols.

Main experimental protocols Before each trial participants will be asked to avoid any strenuous exercise at least for 72 hours. After 7 days of baseline assessment, participants will come to the laboratory. Each of these trials will be separated by at least 5-7 days. Before and after each protocol blood glucose levels (SBP and DPB) will be measured, as well as RPE, enjoyment, affect, and adverse events using the standardized questionaries and rating scales. Moreover, HR will be measured continuously during each exercise session.

1. Participants will come to the laboratory three times a day and the protocols will not last longer than half an hour. Therefore, after a short-term warm-up on the cycle ergometer (5 minutes, the intensity was determined by the participants themselves), short-term, intense bouts of cycling 6x1 minute at 90% HR max with a minute of active break between bouts will be performed (at 50 W). Recovery will last 3 minutes, also at the self-paced. The whole process will be repeated two more times during the day with intervals of 1-4 hours
2. For the SS group, training will consist of three separate sprints on the cycle ergometer separated by 1-4 h. The SS exercise bouts will consist of a 2-minute warm-up followed by a 20-s sprint and then a 1-minute cooldown (three separate workout sessions each lasting 3 min 20 s). The warm-up, cooldown, and recovery periods will all be performed at 50 W. Each sprint will be performed at a resistance of 0.21 N m/kg and include a 10-s period when participants will be advised to accelerate the number of rpm as fast as possible.
3. Control - During CON, participants will come to the lab and remain sedentary throughout this entire period.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years old patients who have been diagnosed with Type 2 diabetes at least 3 months prior to the start of the study according to standard criteria
* BMI between 25 and 35 kg/m2 Inactive patients according to the International Physical Activity Questionnaire
* patients receiving medical therapy (no more than two medications) and not undergoing exogenous insulin therapy
* patients free of injuries and without any contraindications to exercise or chronic diseases that might be disruptive with vigorous activity
* patients should be stable on their current diabetes medications, with no recent changes in their treatment regimen

Exclusion Criteria:

* patients undergoing exogenous insulin therapy or/and receiving more than two glucose-lowering medicaments
* highly physically active on the International Physical Activity Questionnaire (IPAQ)
* patients suffering from any of the ''end-stage'' chronic diseases including: renal disease, liver disease, neuropathy, cardiovascular diseases uncontrolled hypertension
* patients who are strictly prohibited by medical professionals from engaging in vigorous exercise

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-20 (Estimated); Primary Completion 2024-02-20 (Estimated); Study Completion 2024-03-15 (Estimated)

PRIMARY OUTCOMES:
Mean 24-hour blood glucose levels | At baseline (visit 1, week 1) and through main experimental period (visit 5 , week 2, visit 6 - week 3 and visit 7 - week 4).
  Blood glucose levels (mmol/L) will be measured continuously using continuous glucose monitoring system under free-living conditions without providing standardized meals
Time spent in hyperglycemia | At baseline (visit 1, week 1) and through main experimental period (visit 5 , week 2, visit 6 - week 3 and visit 7 - week 4).
  The % of the day spent above 10 mmol/L within 24 hours will be calculated using continuous glucose monitoring system under free-living conditions without providing standardized meals.
Glycemic variability | At baseline (visit 1, week 1) and through main experimental period (visit 5 , week 2, visit 6 - week 3 and visit 7 - week 4).
  Glycemic variability will be measured using the mean amplitude of glycemic excursions (MAGE) and standard deviation (SD) from mean glucose.
Incremental Area Under the Curve (AUC) | At baseline (visit 1, week 1) and through main experimental period (visit 5 , week 2, visit 6 - week 3 and visit 7 - week 4).
  The incremental area under the curve for the glucose response will be calculated using trapezoidal model.

SECONDARY OUTCOMES:
Ratings of perceived exertion (RPE) | RPE will be examined before and after each exercise session during main experimental period.
  RPE will be examined using Borg Scale (0-10 scale) with 1 being ,,very light'' and 10 being ''maximum effort''.
Adverse events | Adverse events will be assessed through main experimental period (visit 5 , week 2; visit 6 - week 3; visit 7 - week 4)
  Adverse events will be evaluated and classified into four different categories: 1) minor and temporary, 2) serious symptoms (potential risk of severe injury or life threatening, 3) manifest injury or disease and 4) death. An adverse event rate will be calculated for each participant as the total number of sessions during which any adverse events occurred divided by the total number of attended sessions.
Exercise enjoyment | Will be assessed immediately after each exercise session during main experimental period.
  The Physical Activity Enjoyment Scale (PACES) will be used to determine the perceived enjoyment after each exercise session. The PACES is an 18-item physical activity/exercise enjoyment scale in which participants are asked to rate "how you feel at the moment about the physical activity/exercise you have been doing" on a 7-point bipolar Likert scale with a total score of 126. Higher scores indicate greater levels of the exercise enjoyment.
Changes in positive and negative affect | Changes in positive and negative affect will be measured before and after each exercise session during main experimental period.
  Changes in positive and negative affect as a result of the exercise bouts will be measured using the positive and negative affect scale (PANAS). The PANAS consists of 20 items, with 10 items measuring positive affect and 10 items measuring negative affect on a 5-point Likert scale. Higher scores indicate higher levels of positive affect.
Blood pressure | SBP and DBP will be measured at baseline before and after each exercise session during main experimental period.
  Both systolic (SBP) and diastolic blood pressure (DBP) will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Milica Pesic, PhD, Study Director — Medical Faculty, University of Nis

REFERENCES:
- [Derived] Lazic A, Dankovic G, Korobeinikov G, Cadenas-Sanchez C, Trajkovic N. Acute effects of different "exercise snacking'' modalities on glycemic control in patients with type 2 diabetes mellitus (T2DM): study protocol for a randomized controlled trial. BMC Public Health. 2025 Feb 11;25(1):566. doi: 10.1186/s12889-025-21669-9. PMID 39934727